CLINICAL TRIAL: NCT04700332
Title: 2-(3-{1-carboxy-5-[(6-18F-fluoro-pyridine-3-carbonyl)-Amino]-Pentyl}-Ureido)-Pentanedioic Acid (PyL) in Patients With High Risk and Biochemically Recurrent Prostate Cancer
Brief Title: PyL in Patients With High Risk and Biochemically Recurrent Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Gary Ulaner, Director Molecular Imaging and Therapy, Hoag Memorial Hospital Presbyterian
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 184-20-CA
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; DCFPyL PET/CT; Staging; Biochemical relapse
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High risk prostate cancer (Experimental): DCFPyL PET/CT will be compared to CT/bone scan for detection of unsuspected metastases in patients with high risk prostate cancer and planned prostatectomy or or radiation therapy
  Interventions: Drug: DCFPyL PET/CT
- Biochemically recurrent prostate cancer (Experimental): DCFPyL PET/CT will be utilized for detection of unsuspected metastases in patients with biochemically recurrent prostate cancer, but with no evidence of disease on CT/bone scan.
  Interventions: Drug: DCFPyL PET/CT

INTERVENTIONS:
Drug: DCFPyL PET/CT — Prostate Membrane Specific Antigen-specific imaging

SUMMARY:
The standard of care imaging of prostate cancer metastases recommended by the National Comprehensive Cancer Network (NCCN), CT of the chest/abdomen/pelvis and bone scan, may be suboptimal. PyL is a novel PET tracer designed to detect prostate specific membrane antigen (PSMA) expressed on prostate cancer cells. PyL PET/CT may provide improved evaluation of clinically significant metastases in patients with prostate cancer.

DETAILED DESCRIPTION:
This will be a phase II clinical trial to assess the clinical value of PyL for detection of disease in pateints with:

1. High risk prostate cancer and planned prostatectomy or radiation therapy (arm 1) and
2. Biochemically recurrent prostate cancer (arm 2) but without evidence of disease of standard of care imaging (CT of the chest/abdomen/pelvis and bone scan).

In both cohorts, PyL PET/CT will be obtained and evaluated by a nuclear radiologist trained in novel PET radiotracers, including PyL. Lesions suspicious for disease of PyL that were unsuspected on standard of care imaging will be selected for biopsy for pathologic confirmation if feasible . Pathology will be used as the reference standard for confirming malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years of age.
2. Histologically confirmed adenocarcinoma of the prostate
3. Patients meet one of the follow criteria:

Cohort 1: High risk prostate cancer (PSA >10, Gleason 8-10, or clinical stage >T2c) and planned prostatectomy or radiation therapy or Cohort 2: Biochemical prostate cancer relapse (Prostate Specific Antigen (PSA) > 0.2 ng/ml in patients following prostatectomy or ≥ 2 ng/ml more than the PSA nadir in patient following radiotherapy, as defined by the ASTRO-Phoenix criteria [18] and no evidence of malignancy on standard of care imaging for metastases (CT of the chest/abdomen/pelvis and bone scan) within 3 months.

Exclusion Criteria:

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
2. Patients who cannot undergo PET/CT scanning because of weight limits. PET/CT scanners may not be able to function with patients over 450 pounds.
3. Change in therapy since standard of care imaging

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Detection of unsuspected metastases in high risk prostate cancer | up to 4 weeks
  Determine the rate of detection of unsuspected metastases in patients with high risk prostate cancer and planned prostatectomy or radiation therapy.
Detection of unsuspected metastases in biochemically recurrent prostate cancer | up to 4 weeks
  Determine the rate of detection of unsuspected metastases in patients with biochemically recurrent prostate cancer, yet no evidence of disease on CT/bone scan.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Fridman, PsyD, RN, Study Director — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Memorial Hospital Presbyterian, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulaner GA, Thomsen B, Bassett J, Torrey R, Cox C, Lin K, Patel T, Techasith T, Mauguen A, Rowe SP, Lindenberg L, Mena E, Choyke P, Yoshida J. 18F-DCFPyL PET/CT for Initially Diagnosed and Biochemically Recurrent Prostate Cancer: Prospective Trial with Pathologic Confirmation. Radiology. 2022 Nov;305(2):419-428. doi: 10.1148/radiol.220218. Epub 2022 Jul 19. PMID 35852431